CLINICAL TRIAL: NCT04416802
Title: A Clinical Study of the Combined Treatment of Platelet-rich Plasma and Low-intensity Extracorporeal Shockwave Therapy on Erectile Dysfunction
Brief Title: Combined Treatment of Platelet-rich Plasma (PRP) and Low-intensity Extracorporeal Shockwave Therapy (Li-ESWT) on Erectile Dysfunction (ED)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ming-Che Liu, MD, Director of Clinical Research Center, Taipei Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N201907013
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Erectile Dysfunction
Keywords: erectile dysfunction; platelet-rich plasma; low-intensity extracorporeal shockwave therapy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP and Li-ESWT treatment (Experimental): Participants diagnosed with erectile dysfunction will receive the combined treatment of platelet-rich plasma and low-intensity extracorporeal shockwave therapy.
  Interventions: Combination Product: autologous platelet-rich plasma and low-intensity extracorporeal shockwave therapy

INTERVENTIONS:
Combination Product: autologous platelet-rich plasma and low-intensity extracorporeal shockwave therapy — The patient who encounters sexual dysfunction and visits our Outpatient Department (OPD) could enter this trial if he meets the inclusion criteria and exclusion criteria.
  1. To fill the questionnaires of International index of erectile function (IIEF) and erectile hardness score (EHS) before starting treatment.
  2. Li-ESWT treatment weekly for three weeks and PRP injection at the same day after the last Li-ESWT treatment.
  3. Coming back at the fourth week and check is there any side effect and fill the questionnaires of IIEF and EHS.
  4. Li-ESWT treatment weekly for three weeks starts on fifth week and PRP injection at the same day after the last Li-ESWT treatment.
  5. Coming back at the eighth week and check is there any side effect and fill the questionnaires of IIEF and EHS.
  6. Coming back at the twelfth week and check is there any side effect and fill the questionnaires of IIEF and EHS.

SUMMARY:
The purpose of this clinical study is mainly to use platelet-rich plasma combined with low-intensity extracorporeal shockwave therapy to treat patients with erectile dysfunction and observe the improvement results.

DETAILED DESCRIPTION:
According to statistics from the Taiwan Society of Andrology, 18 to 25 years old male population in Taiwan having erectile dysfunction (ED) trouble is as high as 5 to 10 percent. At the same time, statistics from the Taiwan Sexual Dysfunction Counseling Training Committee show that as many as 50 percent of men between 40 and 70 years old have erectile dysfunction. Erectile dysfunction is the most common sexual dysfunction in men and is believed to be related to nerve or blood vessel damage, and often significantly affects the patients' quality of life.

PRP is the abbreviation of "platelet-rich plasma". It can release growth factors and cytokines in the body to further promote tissue repair. The results of pre-clinical and clinical trials show that PRP can promote the repair of cavernous tissue, protect erection function of nerve, and stimulate the regeneration of nerve.

Low-intensity extracorporeal shockwave therapy (Li-ESWT) is a non-invasive treatment. Under this treatment, it will help body producing angiogenesis-related proteins, stimulating the formation of small blood vessels, generating new blood vessels at the site to be treated, and increasing the perfusion flow of local tissues. Li-ESWT has been clinically shown to have a significant effect on erectile dysfunction.

The purpose of this clinical study is mainly to use platelet-rich plasma combined with low-intensity extracorporeal shockwave therapy to treat patients with erectile dysfunction and observe the improvement results.

ELIGIBILITY:
Inclusion Criteria:

* Impotence for more than three months
* International index of erectile function, (IIEF) less than 21( including 21)
* Erectile hardness score, (EHS) less than 3( including 3)
* Age over 30 years old

Exclusion Criteria:

* Hypogonadism
* Bleeding tendency
* Could not cooperate with the treatment
* AIDS, syphilis and condyloma victim
* Received radical prostatectomy
* Prostate cancer or pelvis malignant tumor victim
* Gonad dysfunction
* Penis deformities
* Penile prosthesis implantation
* Psychiatric disease victim
* Neural disease ( multiple myeloma , brain atrophy, etc)
* Pacemaker implantation
* Not suitable join this trial judged by Investigator
* Alcohol or drug abuse

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-28 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The Change in Erectile Function | Baseline, the 4th week, 8th week, and 12th weeks
  Using the International Index of Erectile Function (IIEF) questionnaire.
The Change in Erectile Function | Baseline, the 4th week, 8th week, and 12th weeks
  Using the Erectile Hardness Scale (EHS) questionnaire to evaluate the efficacy of combined treatment of PRP and Li-ESWT

SECONDARY OUTCOMES:
Incidents of Side Effects | the 4th week, 8th week, and 12th weeks
  To observe whether there are side effects

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Che Liu, MD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanderson LM, Bryant A. Effectiveness and safety of prolotherapy injections for management of lower limb tendinopathy and fasciopathy: a systematic review. J Foot Ankle Res. 2015 Oct 20;8:57. doi: 10.1186/s13047-015-0114-5. eCollection 2015. PMID 26500703
- [Background] Rosenthal AR, Harbury C, Egbert PR, Rubenstein E. Use of a platelet-fibrinogen-thrombin mixture as a corneal adhesive: experiments with sutureless lamellar keratoplasty in the rabbit. Invest Ophthalmol. 1975 Nov;14(11):872-5. PMID 1102485
- [Background] Wu YN, Wu CC, Sheu MT, Chen KC, Ho HO, Chiang HS. Optimization of platelet-rich plasma and its effects on the recovery of erectile function after bilateral cavernous nerve injury in a rat model. J Tissue Eng Regen Med. 2016 Oct;10(10):E294-E304. doi: 10.1002/term.1806. Epub 2013 Aug 16. PMID 23950105
- [Background] Wu CC, Wu YN, Ho HO, Chen KC, Sheu MT, Chiang HS. The neuroprotective effect of platelet-rich plasma on erectile function in bilateral cavernous nerve injury rat model. J Sex Med. 2012 Nov;9(11):2838-48. doi: 10.1111/j.1743-6109.2012.02881.x. Epub 2012 Aug 20. PMID 22906160
- [Background] Ruan Y, Zhou J, Kang N, Reed-Maldonado AB, Tamaddon A, Wang B, Wang HS, Wang G, Banie L, Lin G, Liu J, Lue TF. The effect of low-intensity extracorporeal shockwave therapy in an obesity-associated erectile dysfunction rat model. BJU Int. 2018 Jul;122(1):133-142. doi: 10.1111/bju.14202. Epub 2018 Apr 17. PMID 29573106
- [Background] Scott S, Roberts M, Chung E. Platelet-Rich Plasma and Treatment of Erectile Dysfunction: Critical Review of Literature and Global Trends in Platelet-Rich Plasma Clinics. Sex Med Rev. 2019 Apr;7(2):306-312. doi: 10.1016/j.sxmr.2018.12.006. Epub 2019 Mar 2. PMID 30833169
- [Background] Dong L, Chang D, Zhang X, Li J, Yang F, Tan K, Yang Y, Yong S, Yu X. Effect of Low-Intensity Extracorporeal Shock Wave on the Treatment of Erectile Dysfunction: A Systematic Review and Meta-Analysis. Am J Mens Health. 2019 Mar-Apr;13(2):1557988319846749. doi: 10.1177/1557988319846749. PMID 31027441
- [Background] Patel P, Huang C, Molina M, Ramasamy R. Clinical trial update on shockwave therapy and future of erectile function restoration. Int J Impot Res. 2019 May;31(3):206-208. doi: 10.1038/s41443-019-0115-1. Epub 2019 Jan 22. PMID 30670840